CLINICAL TRIAL: NCT06554782
Title: Children's Compliance With Toothbrushing Using Manual U-shaped Toothbrush Versus Regular Manual Toothbrush
Brief Title: Children's Compliance With Toothbrushing Using Manual U-shaped Toothbrush Versus Regular Toothbrush
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Sobhy Saeed, master degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: U-shaped toothbrush
Record Dates: First submitted 2024-08-02; First posted 2024-08-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Manual Toothbrush

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual u-shaped toothbrush (Experimental): manual u-shaped toothbrush with arm angled 45 degrees to brush upper and lower arch at the same time
  Interventions: Device: manual u-shaped toothbrush
- manual toothbrush (Experimental): manual toothbrush with soft bristles and circular movement to clean each quadrant separately
  Interventions: Device: manual u-shaped toothbrush

INTERVENTIONS:
Device: manual u-shaped toothbrush — manual u-shaped toothbrush with bristles angled 45 degrees to brush upper and lower teeth at the same time

SUMMARY:
To assess the child's compliance towards manual U-shaped toothbrush versus regular manual toothbrush.

DETAILED DESCRIPTION:
Research has shown that an undesirably high proportion of communities find thorough toothbrushing with a standard manual toothbrush challenging to achieve a plaque-free state, as evidenced by high worldwide gingivitis and periodontitis. This is consistent with investigations that reveal insufficient frequency of brushing, poor brushing technique, and inadequate brushing session duration when compared with standard-of-care professional recommendations.

The U-shaped brush is an intervention chosen for the present study because it can attract children's attention and make brushing fun and routine. With bristles angled at 45° and available in various sizes according to age, the U-shaped brush is useful for removing plaque. It can be used starting at age three or older. It is dependable for children because its two-sided design can clean the upper and lower arches in one motion. Since design affects plaque removal to varying degrees, various authors have examined the effects of different toothbrush designs on plaque removal.

ELIGIBILITY:
Inclusion Criteria:

1. children aged 5 to 10 years, in good general health, and medically free.
2. Cooperative patients who will comply with follow-ups.
3. Parents who accept to sign informed consent.

Exclusion Criteria:

1. Children with fixed or removable orthodontic appliances.
2. Children with a physical disability, and medical disability.
3. Children who will be unable to attend follow-up visits.
4. Parents refuse to give written formed consent.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
compliance of patient | 1 week
  questioning the parents about compliance either yes or no

SECONDARY OUTCOMES:
full mouth plaque score | 1 week
  Turesky modified Quigley-Hein plaque index technique index score: total score/number of surfaces examined 0-1= low >2= high

CONTACTS AND LOCATIONS:
Overall Officials: Randa Youssef AbdelGawad, professor, Study Director — Cairo University; Rana Tarek Bartaw, assistant professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashkenazi M, Bidoosi M, Levin L. Factors associated with reduced compliance of children to dental preventive measures. Odontology. 2012 Jul;100(2):241-8. doi: 10.1007/s10266-011-0034-1. Epub 2011 Jun 23. PMID 21698350
- [Result] Davidovich E, Ccahuana-Vasquez RA, Timm H, Grender J, Cunningham P, Zini A. Randomised clinical study of plaque removal efficacy of a power toothbrush in a paediatric population. Int J Paediatr Dent. 2017 Nov;27(6):558-567. doi: 10.1111/ipd.12298. Epub 2017 May 11. PMID 28494116